CLINICAL TRIAL: NCT07131956
Title: Immune Biomarkers in Prostate Cancer Patients Treated With Brachytherapy (ImmunBioProBrachy)
Brief Title: Immune Biomarkers in Prostate Cancer Patients Treated With Brachytherapy
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Bavarian Cancer Research Center (BZKF) (Unknown); University Hospital Augsburg (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Claudia Schweizer, Claudia Schweizer MD, University of Erlangen-Nürnberg Medical School
Other Study IDs: ImmunBioProBrachy
Record Dates: First submitted 2025-08-03; First posted 2025-08-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer (Diagnosis); Prostate Cancer Patients Who Have Brachytherapy Seed Implant; Prostate Cancer Patients Treated by Radiotherapy; Prostate Cancer Recurrent
Keywords: Immune-profiling in prostate cancer patients; brachytherapy for prostate cancer; interstitial brachytherapy for prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — wohle blood, prostate tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary brachytherapy: Patients receiving sole primary brachytherapy (either LDR-BT or HDR-BT) for low or low intermediate risk prostate cancer
- Salvage brachytherapy: Patients receiving sole brachytherapy (either PDR-BT or HDR-BT) for locally recurrent prostate cancer after prior irradiation with prostate in situ

SUMMARY:
Analysis of peripheral immune cells before, during, and after brachytherapy treatment. Corresponding analysis of tissue samples collected during brachytherapy treatment.

ELIGIBILITY:
Inclusion Criteria Arm 1:

* Primary treatment with I-125 seeds or HDR-BT
* No previous treatment for prostate cancer
* Age ≥ 18 years

Inclusion Criteria Arm 2:

* HDR- or PDR-BT
* No radiation therapy within three months before salvage treatment
* Complete documentation available on previous treatment for prostate cancer
* No history of prostatectomy
* Age ≥ 18 years

Exclusion Criteria:

* Pre-existent auto-immune disease
* patients under bloodthinning medication
* substance abuse

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients planning to undergo sole brachytherapy treatment
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal changes of peripheral immune cells and cell-free DNA and tumor-associated tissue in patients with prostate cancer treated with brachytherapy | Blood withdrawal pre-brachytherapy treatment, during surgery, one day after brachytherapy and at the first follow-up visit 4-12 weeks later. Tissue samples at every brachytherapy procedure.
  Longitudinal changes of peripheral immune cells and cell-free DNA and tumor-associated tissue in patients with prostate cancer treated with brachytherapy in the primary as well as in the recurrent setting.

SECONDARY OUTCOMES:
Treatment-related toxicity | Up to 6 months
  Acute toxicity related to brachytherapy
recurrence-free survival | Up to 6 months
  recurrence-free survival
Overall survival | Up to 6 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Schweizer, MD, Principal Investigator — Strahlenklinik Universitätsklinikum Erlangen; Anna-Jasmina Donaubauer, Dr. rer. nat., Principal Investigator — Strahlenklinik Universitätsklinikum Erlangen
Locations (3):
- Germany (3):
  - Klinik für Strahlentherapie, Augsburg, Bavaria
  - Strahlenklinik Erlangen, Erlangen, Bavaria
  - Klinik und Poliklinik für Strahlentherapie und Radioonkologie, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: No